CLINICAL TRIAL: NCT00364390
Title: A Phase I Open Label Pilot Study to Evaluate the Safety, Efficacy and Tolerability of Anginera for Adults With Left Ventricular Dysfunction AND Reversible Myocardial Ischemia Undergoing CABG Surgery
Brief Title: A Study of Anginera In Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theregen, Inc. (Industry)
Responsible Party: Gary Gentzkow, M.D. Chief Medical Officer, Theregen, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITT-101
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease
Keywords: CABG; Anginera; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Anginera, a human tissue replacement therapy

SUMMARY:
This is a first in man, Phase I safety study of Anginera in adults with Left Ventricular Dysfunction (LVD) and Reversible Myocardial Ischemia undergoing a CABG procedure.

DETAILED DESCRIPTION:
A prospective, multicenter, open-label Phase I safety study of Anginera. Adults with Left Ventricular Dysfunction and reversible myocardial ischemia who are undergoing a CABG procedure, who have at least one graftable vessel and at least one coronary vessel not amenable to bypass or PCI (Percutaneous Coronary Intervention)will be recruited. Three pieces of Anginera will be placed on the area of the surface of the ventricle, including the area supplied by the vessel or vessels that cannot be bypassed, as well as surrounding myocardium. Patients will be followed for 12 months after the surgery at which Anginera is implanted.

The primary objective is to determine safety. The secondary objectives are to determine regional myocardial perfusion and regional left ventricular performance and to investigate the utility of measures of patient perception of improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been referred for CABG
* Left ventricular ejection fraction (LVEF) greater than 20%
* Patients have CAD involving at least two (2) coronary arteries, with at least one or more vessel(s) having disease not amenable to bypass grafting or PCI
* There is a region of myocardium served by the vessel(s) defined above that has objective evidence of multi-distribution reversible ischemia based on a 17-segment assessment of reversible defects on SPECT/Thallium.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Patient undergoing valve replacement or valve modification
2. Patient with significant or malignant ventricular arrhythmias, defined as a patient being treated for ventricular tachycardia and/or ventricular fibrillation with an implantable cardioverter/defibrillator (ICD) or a patient being treated with Amiodarone for these same tachyarrhythmias. (Note: having an implantable cardioverter/defibrillator (ICD) per se, in a patient who does not have significant or malignant ventricular arrhythmias, does not exclude the patient from this study.)
3. Patient requires urgent coronary artery bypass surgery

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Physical exam and interval medical history
CBC and differential
Serum cardiac markers-Troponin I
Serum chemistries and urinalysis
Resting electrocardiogram (ECG)
24 hour Holter monitor
Adverse Events reporting

CONTACTS AND LOCATIONS:
Overall Officials: Bartley P Griffith, MD, Principal Investigator — University of Maryland, Baltimore; George Tellides, M.D., Ph.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University School of Medicine,, New Haven, Connecticut
  - University of Maryland School of Medicine, Baltimore, Maryland